CLINICAL TRIAL: NCT03886792
Title: A Home-Based Biofeedback Program to Augment Recovery After Perinatal Brachial Plexus Injury
Brief Title: Brachial Plexus Birth Palsy: Reinforcement Paradigm to Augment Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chapman University (Other)
Collaborators: American Society for Surgery of the Hand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1408
Record Dates: First submitted 2019-02-25; First posted 2019-03-22 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Brachial Plexus Palsy
MeSH Terms: interventions — Drug Interactions

STUDY DESIGN:
Intervention Model Description: Feasibility Randomized Controlled Trial with one experimental and one control group
Who Masked: Outcomes Assessor
Masking Description: Blind to treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triggered Reinforcement (Experimental): This group will participate in a home-based experimental intervention for 10 minutes, twice/day for 10 days within 2 weeks. The infants will be supported in sitting with a tray secured anterior to the trunk. This intervention will involve reinforcement of biceps muscle activation in the affected arm if the infant generates a muscle contraction above a pre-set threshold (V). The threshold needed to trigger a toy to move and make sounds (reinforcement) will be set at baseline as determined by surface electromyography (SEMG). During the training time-points, the parent or care-giver will be allowed to sing or talk to the infant but are not to shake the toys or place dowel-based rattles or toys in either palm of the infant.
  Interventions: Behavioral: Triggered reinforcement
- Social Interaction (Sham Comparator): This group will participate in a home-based dose-equivalent control intervention for 10 minutes, twice/day for 10 days within 2 weeks. The infants will be supported in sitting with a tray. This control program will combine social interaction between infant/parent with the opportunity for self-initiated play with toys repeatedly placed on the tray. A toy will be placed in front of the infant seat and tray but it will not be connected to the SEMG unit nor will the infant have an SEMG electrode attached over the biceps. During the intervention, the parent or care-giver will be allowed to sing or talk to the infant but are not to shake the toys or place dowel-based rattles or toys in either palm of the infant.
  Interventions: Behavioral: Social interaction

INTERVENTIONS:
Behavioral: Triggered reinforcement — This group will participate in a home-based experimental intervention for 10 minutes, twice/day for 10 days within 2 weeks. The infants will be supported in sitting with a tray secured anterior to the trunk. This intervention will involve reinforcement of biceps muscle activation in the affected arm if the infant generates a muscle contraction above a pre-set threshold (V). The threshold needed to trigger a toy to move and make sounds (reinforcement) will be set at baseline as determined by surface electromyography (SEMG). During the training time-points, the parent or care-giver will be allowed to sing or talk to the infant but are not to shake the toys or place dowel-based rattles or toys in either palm of the infant.
  Arms: Triggered Reinforcement
Behavioral: Social interaction — This group will participate in a home-based dose-equivalent control intervention for 10 minutes, twice/day for 10 days within 2 weeks. The infants will be supported in sitting with a tray. This control program will combine social interaction between infant/parent with the opportunity for self-initiated play with toys repeatedly placed on the tray. A toy will be placed in front of the infant seat and tray but it will not be connected to the SEMG unit nor will the infant have an SEMG electrode attached over the biceps. During the intervention, the parent or care-giver will be allowed to sing or talk to the infant but are not to shake the toys or place dowel-based rattles or toys in either palm of the infant.
  Arms: Social Interaction

SUMMARY:
Infants who sustain an injury to the brachial plexus in the perinatal period are at high-risk for long-term neuromuscular deficits and prehensile dysfunction. If recovery is delayed because of slow axonal regrowth, disuse atrophy and secondary musculoskeletal deficits may develop. The investigators' hypothesis is that early, intensive intervention designed to foster muscle activation is essential to optimize outcomes after brachial plexus injury and may supplement rehabilitation and microsurgery. This proposal targets infants who are non-surgical candidates. Yet, future studies will examine whether the investigators' experimental intervention can hasten recovery from microsurgery and will examine which post-operative time-point is best to employ it. The investigators' intervention shows promise to increase muscle activation and improve arm function in infants with brachial plexus birth palsy (BPBP) through contingent reinforcement based on a pilot study.

DETAILED DESCRIPTION:
The investigator's study objectives are to (1) test the feasibility of a parent-lead in-home 2-week intervention for infants with BPBP; and (2) determine the effect size for the primary outcome measure(s) in preparation for a future definitive randomized controlled trial (RCT). In this feasibility RCT, the investigators will compare two in-home interventions in 3 to 12-month-old infants with upper trunk BPBP; n=12 per group: (1) experimental; and (2) dose-equivalent active control. For the experimental intervention, infants will trigger a musical toy to move and play via biceps contraction above a preset individual threshold. For the control intervention, toys will be available to play with, yet, there will be no reinforcement for biceps activation.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 3 to 12 months with upper trunk brachial plexus birth palsy confirmed by an attending Hand and Upper Extremity Surgeon;
2. Full-term at birth;
3. A minimum score of '1' (0-7 scale) in elbow flexion of affected arm (isometric contraction) based on the Active Movement Scale (AMS);
4. Score ≥ 25th percentile on the motor subtest of the Bayley Scales of Infant and Toddler Development, 3rd Edition (BSITD-III®);
5. Ability to sustain attention/arousal for a 10 minute training period based on criteria from the Neonatal Behavioral Assessment for an awake-alert state.

Exclusion Criteria:

1. Visual/auditory deficits;
2. Nerve repair/shoulder surgery;
3. Excessive crying during session(s);
4. Shoulder, elbow, or wrist joint contractures > 20° in the affected arm;
5. An inability to trigger the musical-toy to play at baseline.

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the integral of biceps brachii muscle activation post-intervention | Baseline, Immediately post-intervention, 1-month post-intervention, 3-months post-intervention
  Change in the magnitude of biceps muscle activation (Volts x time) post-intervention

SECONDARY OUTCOMES:
Change in day-long arm activity based on the resultant acceleration (ms*m/s2) | Baseline, Immediately post-intervention, 1-month post-intervention, 3-months post-intervention
  Resultant acceleration of arm activity (ms*m/s2) over one daytime period
Parent Perception Questionnaire to examine feasibility of parent-run intervention - self designed | Immediately post-intervention
  Parent Perception Questionnaire with responses based on short-answer and a 5-point Likert scale. The Likert scale will measure responses on a 1-5 range with lower scores indicating a better outcome. A frequency distribution will be used to represent the responses on each Likert subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Susan V Duff, EdD,PTOT,CHT, Principal Investigator — Chapman University
Locations (1):
- Children's Hospital of Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Duff SV, Sargent B, Kutch JJ, Berggren J, Leiby BE, Fetters L. Using Contingent Reinforcement to Augment Muscle Activation After Perinatal Brachial Plexus Injury: A Pilot Study. Phys Occup Ther Pediatr. 2017 Oct 20;37(5):555-565. doi: 10.1080/01942638.2017.1290733. Epub 2017 Apr 20. PMID 28426263
- [Result] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. Pilot Feasibility Stud. 2016 Oct 21;2:64. doi: 10.1186/s40814-016-0105-8. eCollection 2016. PMID 27965879
- [Result] Foad SL, Mehlman CT, Ying J. The epidemiology of neonatal brachial plexus palsy in the United States. J Bone Joint Surg Am. 2008 Jun;90(6):1258-64. doi: 10.2106/JBJS.G.00853. PMID 18519319
- [Result] Sullivan GM, Artino AR Jr. Analyzing and interpreting data from likert-type scales. J Grad Med Educ. 2013 Dec;5(4):541-2. doi: 10.4300/JGME-5-4-18. No abstract available. PMID 24454995